CLINICAL TRIAL: NCT06856837
Title: - IKF/AIO-QUINTIS - A Randomized Phase II Trial Evaluating Fruquintinib in Combination With Tislelizumab in Microsatellite Stable / Proficient Mismatch Repair (MSS/pMMR) Metastatic Colorectal Cancer Without Active Liver Metastases
Brief Title: - IKF/AIO-QUINTIS - Evaluating Fruquintinib in Combination With Tislelizumab in Microsatellite Stable / Proficient Mismatch Repair (MSS/pMMR) Metastatic Colorectal Cancer Without Active Liver Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUINTIS
Record Dates: First submitted 2025-02-18; First posted 2025-03-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; tislelizumab; trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Participants eligible for this trial will be randomized 1:1 into one of the two arms (experimental Arm A and control Arm B) stratified by: I) Previous anti-angiogenic therapy (yes vs. no), II) BRAF/RAS mutation status (wildtype vs. mutation), III) History of liver metastases (never vs. prior but treated)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): * Fruquintinib (orally, 5 mg once a day, at day 1-21 of each 28-day cycle [Q4W]) plus
  * Tislelizumab (i.v., 400 mg, at day 1 of each 42-day cycle [Q6W])
  Interventions: Drug: Fruquintinib; Drug: Tislelizumab
- Arm B (Active Comparator): * Trifluridine/tipiracil (orally, 35 mg/m2 twice a day, day 1-5 and day 8-12 of each 28-day cycle [Q4W]) plus
  * Bevacizumab (i.v., 5 mg/kg, at day 1 of each 14-day cycle [Q2W])
  Interventions: Drug: Trifluridine/tipiracil; Drug: Bevacizumab

INTERVENTIONS:
Drug: Fruquintinib — highly selective and potent oral inhibitor of vascular endothelial growth factor receptors (VEGFRs) 1, 2, and 3
  Other Names: Fruzaqla
  Arms: Arm A
Drug: Tislelizumab — humanized immunoglobulin G4 (IgG4)-variant monoclonal antibody (mAb) against human programmed cell death-1 (PD-1)
  Other Names: Tevimbra
  Arms: Arm A
Drug: Trifluridine/tipiracil — trifluridine, a nucleoside analog, and tipiracil, a thymidine phosphorylase inhibitor
  Other Names: Lonsurf
  Arms: Arm B
Drug: Bevacizumab — recombinant humanized anti-VEGF monoclonal antibody composed of human IgG1 framework regions and antigen-binding, complementarity-determining regions from a murine monoclonal antibody (muMAb VEGF A4.6.1)
  Other Names: Avastin
  Arms: Arm B

SUMMARY:
This is a prospective, randomized, open-label, multicenter phase II investigating the therapy of Fruquintinib in combination with Tislelizumab in patients with MSS/pMMR metastatic colorectal cancer without liver metastases.

DETAILED DESCRIPTION:
Participants eligible for this trial will be randomized 1:1 into one of the two arms (Arm A and Arm B) stratified by: I) -Previous anti-angiogenic therapy (yes vs. no), II) BRAF/RAS mutation status (wildtype vs. mutation) or III) History of liver metastases (never vs. prior but treated).

Patients in Arm A (experimental arm) will receive Fruquintinib (orally, 5 mg once a day, at day 1-21 of each 28-day cycle [Q4W]) plus Tislelizumab (i.v., 400 mg, at day 1 of each 42-day cycle [Q6W]).

Patients in Arm B (control arm) will receive Trifluridine/tipiracil (orally, 35 mg/m2 twice a day, day 1-5 and day 8-12 of each 28-day cycle [Q4W]) plus Bevacizumab (i.v., 5 mg/kg, at day 1 of each 14-day cycle [Q2W]).

The treatment will be performed until disease progression, unacceptable toxicity, patients' request, or end of protocol-defined treatment time (maximum of 15 months).

All patients will be followed up for a maximum of 18 months after last patient in or until death, withdrawal of consent or loss to follow-up, whatever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Patient* provide signed informed consent form.
2. Patient is ≥ 18 years at the time of given informed consent.
3. Patient has been diagnosed with histologically or cytologically proven microsatellite stable (MSS)/proficient mismatch repair (pMMR) metastatic adenocarcinoma of the colon or rectum, which is not amenable to potentially curative resection.
4. Known RAS (KRAS or NRAS) and BRAF V600E mutational status. Note: These mutations are mutually exclusive. Therefore, if one of the factors is mutated, it is not required to determine the mutation status of the others, as they are then assumed to be wildtype.
5. Patient without liver metastases (NLM) defined as subjects without active liver metastases at screening as determined on baseline imaging of the liver as performed by CT scan with contrast or MRI. Definitively treated liver metastases (which includes surgical resection, microwave or radiofrequency ablation, or stereotactic body radiation therapy, but not yttrium-90 or chemoembolization alone) that were treated at least 3 months prior to enrollment with no evidence of radiologic progression on subsequent imaging are considered to be non-active liver metastases.
6. Patient received at least one line of previous treatment with a fluoropyrimidine, oxaliplatin, irinotecan, VEGF(R) and if indicated EGFR and/or BRAF inhibitors in the advanced setting, or the patient has been intolerable or ineligible to those treatments.
7. Patient has an ECOG performance status ≤ 1.
8. Patient has a life expectancy > 16 weeks.
9. Patient has adequate hematological, hepatic and renal function.

   1. Absolute number of neutrophils (ANC) ≥ 1.5 x 109/L
   2. Platelets ≥ 100 x 109/L
   3. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) (or < 2 x ULN in case of prior liver involvement or Gilbert's disease)
   4. AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN, AP ≤ 5 x ULN
   5. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (measured by 24 h urine) ≥ 30 mL/min (i.e., if serum creatinine level is > 1.5 x ULN, then a 24-hour urine test must be performed to check the creatinine clearance to be determined).
   6. Urinary protein ≤2+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥3+, a 24-hour urine collection for protein must demonstrate <2000 mg of protein in 24 hours to allow participation in this protocol)
10. Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy).
11. Female patients of childbearing potential or male patients in Arm B with female partners of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 6 months after the last trial treatment. Male patients in Arm B with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy. Female patients of child-bearing potential must have a negative pregnancy test within the last 7 days prior to the start of trial therapy.
12. Patient is willing and able to comply with the protocol (including contraceptive measures) for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

    * There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the trial gender-independently.

Exclusion Criteria:

1. Patient has known allergic / hypersensitive reactions to at least one of the treatment components
2. Patient had previous malignancy other than that under study within 3 years or concomitant malignancy, except: those with a 5-year overall survival rate of more than 90%, e.g. non-melanomatous skin cancer or adequately treated in situ cervical cancer
3. Patient received previous treatment with Fruquintinib, trifluridine/tipiracil, regorafenib or an anti-PD-1/anti-PD-L1 antibodies.
4. Patient receives current treatment with any anti-cancer therapy, such as systemic immunotherapy, chemotherapy, or hormone therapy within ≤ 2 weeks prior to study treatment start.
5. Patient receives simultaneous treatment with a different anti-cancer therapy other than that provided for in the trial (excluding palliative radiotherapy for symptom control).
6. Patient has known untreated or symptomatic CNS or leptomeningeal metastases.
7. Patient has impaired cardiac function or clinically significant cardiac disease including unstable angina within 6 months before the first dose of study treatment, acute myocardial infarction < 6 months prior to the first dose of study treatment, New York Heart Association (NYHA) class II-IV congestive heart failure, uncontrolled hypertension (defined as an average systolic blood pressure > 160 mmHg or diastolic > 100 mmHg despite optimal treatment, uncontrolled cardiac arrhythmias requiring antiarrhythmic therapy other than beta blockers or digoxin, active coronary artery disease or corrected QT interval (QTc) ≥ 470.
8. Patient has history of uncontrolled infection with human deficiency virus (HIV) or chronic infection with hepatitis B or C virus (HBV, HCV).
9. Patient has evidence of bleeding diathesis.
10. Patient has history of gastrointestinal perforation or fistulae in past 6 months or risk factors for perforation.
11. Patient has grade 3-4 gastrointestinal bleeding within 3 months prior to first dose of trial therapy.
12. Use of strong inducers or inhibitors of CYP3A4 within 2 weeks (or 5 half-lives, whichever is longer) before the first dose of study drug (see Appendix 4 for examples).
13. Patient had a major surgery within 2 weeks prior to first dose of trial therapy.
14. Patient experienced severe, life-threatening, or recurrent (Grade 2 or higher) immune-mediated adverse events (AEs) or infusion-related reactions including those that led to permanent discontinuation while on treatment with immune-oncology agents.
15. Patient received prior immunosuppressive therapy: immunosuppressive doses of systemic medications of > 10 mg/day of prednisone or equivalent must be discontinued ≥ 2 weeks before the first dose of study treatment. Short courses of high dose corticosteroids and/or continuous low dose of prednisone (< 10 mg/day) are permitted. In addition, inhaled, intranasal, intraocular, and/or joint injections of corticosteroids are allowed.
16. Patient has active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study.
17. Patient has history of solid organ transplantation .
18. Patient has history of thromboembolic events (including deep vein thrombosis and pulmonary embolism) within the past 6 months or history of stroke and/or transient ischemic attack within the last 12 months.
19. Patients has evidence of any other serious concomitant or medical condition that, in the opinion of the investigator, presents a high risk of complications to the patient or reduces the likelihood of clinical effect.
20. Female patient is pregnant or breast feeding or planning to become pregnant within and up to 6 months after end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of Fruquintinib in combination with the PD-1 inhibitor Tislelizumab in MSS/pMMR metastatic colorectal cancer without liver metastases. | up to 54 month
  Progression-free survival (PFS), defined as time from randomization until date of progression acc. to RECIST v1.1 or death due to any cause.

SECONDARY OUTCOMES:
Overall survival | up to 54 month
  Overall survival (OS), defined as time from randomization until date of death due to any cause.
Objective response rate | up to 54 month
  Objective response rate (ORR), defined as proportion of patients achieving complete or partial response (CR/PR) acc. to RECIST v1.1.
Disease control rate | up to 54 month
  Disease control rate (DCR), defined as proportion of patients achieving CR, PR, or stable disease (SD) acc. to RECIST v1.1.
Duration of response | up to 54 month
  Duration of response (DoR), defined as time from response initiation (when either CR or PR is first determined) to disease progression acc. to RECIST v1.1 or death due to any cause.
To evaluate the safety and tolerability of Fruquintinib in combination with the PD-1 inhibitor Tislelizumab in MSS/pMMR metastatic colorectal cancer without liver metastases. | up to 54 month
  Assessment of safety of the treatment as determined by the incidence, nature, causality, frequency, timing, and severity of adverse events using NCI CTCAE v5.0.
To assess health-related quality of life (HRQoL) data of Fruquintinib in combination with the PD 1 inhibitor Tislelizumab in MSS/pMMR metastatic colorectal cancer without liver metastases. | up to 54 month
  Assessment of HRQoL during treatment and follow-up using EORTC QLQ C30 and EQ-5D-5L questionnaires.

OTHER OUTCOMES:
Exploratory Translational Objectives | up to 54 month
  To correlate analysis between selected blood (such as ctDNA, chemokines/cytokines and metabolites) and stool (microbiota composition and metabolites) parameters and clinical data as well as dietary information to identify molecular biomarkers predictive for tumor response and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Frankfurter Institut für Klinische Krebsforschung IKF GmbH; Alexander Stein, Prof. Dr., Principal Investigator — Hämatologisch-Onkologische Praxis Eppendorf University Cancer Center Hamburg
Locations (23):
- Austria (3):
  - Ordensklinikum Linz GmbH, Linz
  - SCRI CCCIT Ges.m.b.H., Salzburg
  - Noe LGA Gesundheit Thermenregion GmbH, Wiener Neustadt
- Germany (20):
  - Klinikum St. Marien Amberg, Amberg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Charite Universitaetsmedizin Berlin KöR, Berlin
  - HELIOS Emil von Behring Berlin, Berlin
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Universitätsklinikum Düsseldorf Klinik für Gastroenterologie, Hepatologie und Infektiologie Gastroonkologische Studienzentrale, Düsseldorf
  - KEM | Klinik für Internistische Onkologie gGmbH, Essen
  - Universitätsklinikum Essen, Essen
  - Goethe University Frankfurt, Frankfurt
  - Institut für Klinisch-Onkologische Forschung am Krankenhaus Nordwest, Frankfurt am Main
  - Hamburg Hämatologisch-Onkologische Praxis Eppendorf-Facharztzentrum Eppendorf, Hamburg
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Marienhospital Herne, Herne
  - Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - Klinikum der Universität München AöR, München
  - Klinikum rechts der Isar TU München, München
  - Leopoldina Krankenhaus Schweinfurt, Schweinfurt
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No